CLINICAL TRIAL: NCT02213172
Title: Evaluation of the Efficacy of Two Probiotic Strains for Irritable Bowel Syndrome: an 8-Week, Randomized, Placebo-Controlled Study
Brief Title: Evaluation of the Efficacy of Two Probiotic Strains for Irritable Bowel Syndrome
Acronym: 14PIHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 14PIHL
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Probiotic; Constipation; Bifidobacterium longum; Lactobacillus paracasei; Lallemand Health Solutions
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Bifidobacterium longum R0175 (Experimental): 10 x 10^9 CFU per capsule, 1 capsule daily for 8 weeks
  Interventions: Dietary Supplement: Bifidobacterium longum R0175
- Lactobacillus paracasei HA-196 (Experimental): 10 x 10^9 CFU per capsule, 1 capsule daily for 8 weeks
  Interventions: Dietary Supplement: Lactobacillus paracasei HA-196
- Placebo (Placebo Comparator): 1 capsule daily for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum R0175
  Arms: Bifidobacterium longum R0175
Dietary Supplement: Lactobacillus paracasei HA-196
  Arms: Lactobacillus paracasei HA-196
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if two different probiotic strains, Lactobacillus paracasei HA-196 and Bifidobacterium longum R0175, are effective in helping subjects manage the symptoms of IBS

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18 years and older.
* IBS diagnosis according to Rome III criteria and referral to this study by a clinician. That is, recurrent abdominal pain or discomfort (i.e., uncomfortable sensation other than pain) at least 2 days/month in the last 3 months (response to question 1 of the IBS Rome III module questionnaire > 2) associated with 2 or more of the following:

  * Improvement with defecation (response to question 4 of the IBS Rome III module questionnaire > 0);
  * Onset associated with a change in stool frequency (response to question 5 or 6 of the IBS Rome III module questionnaire > 0);
  * Onset associated with a change in stool form (appearance). (response to question 7 or 8 of the IBS Rome III module questionnaire > 0).
* For women, the abdominal pain or discomfort should be experienced during days other than menstrual bleeding (response to question 2 of the IBS Rome III module questionnaire = 0 or 2)
* Criterion must be fulfilled for the last 3 months with symptom onset at least 6 months prior to screening (response to question 3 of the IBS Rome III module questionnaire = 1).
* A copy of the IBS module is provided in Appendix A: IBS Rome III Module Questionnaire
* Participants from the general population who have IBS symptoms, without a previous diagnosis, will be assessed by the Principle Investigator and included in the study if differential diagnosis confirms IBS. The Principle Investigator will confirm the diagnosis of IBS in any potential participants who have a previous diagnosis of IBS.
* Subjects experiencing a pain/discomfort frequency of at least 2 days a week during the run-in period. At visit 2, subjects will be asked "In the last 2 weeks, how often each week did you have discomfort or pain anywhere in your abdomen? ". The answer must be at least 2.
* Subjects diagnosed with IBS who have depression may be included
* Absence of black color (melena) or blood in stools.
* Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits.
* Willingness to discontinue consumption of probiotics (e.g. yogurts, with live, active cultures or supplements).
* Able to provide informed consent.

Exclusion Criteria:

* Subjects with a history of suicidal ideation, or current suicidal ideation
* Previous history of gastrointestinal surgery (except appendectomy, cholecystectomy, hernia repair, or hemorrhoidectomy).
* Other gastrointestinal diseases (except hemorrhoids and uncomplicated diverticula), as assessed by ultrasonography, colonoscopy, or rectoscopy, or history of Clostridium difficile-associated diarrhea.
* A family history (immediate family i.e. siblings and parents) of colorectal cancer, inflammatory bowel disease and/or celiac spruce.
* Co-existing organic gastrointestinal disease.
* Presence of rectal bleeding, recent weight loss (greater than 5 kg in the past month) or iron deficiency anemia.
* History of, or current diagnosis of, liver disease, kidney disease, pulmonary disease, cardiovascular disease, pancreatic disease, any cancer.
* Presence of immune-compromised conditions such as AIDS, lymphoma or undergoing long-term corticosteroid treatment
* Presence or history of neurological disorders, or significant psychiatric illness.
* History of, or current diagnosis of, pelvic floor dyssynergia.
* Positive drug or alcohol screen or recent history of drug or alcohol abuse (within 3 years of screening).
* Milk or soy allergy.
* Use of another investigational product within 3 months of the screening visit. The screened participant could be eligible to participate after a washout period.
* Positive pregnancy test in women of child-bearing potential.
* Pregnant or breast-feeding or planning on becoming pregnant.
* Women of child-bearing potential not using effective contraception. Acceptable methods of birth control include:

  * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
  * Intrauterine devices
  * Vasectomy of partner (shown successful as per appropriate follow-up)
  * Double barrier method (use of physical barrier by both partners)
* Use of any antibiotic drug (e.g., neomycin, rifaximin) within 1 month of screening. The screened participant could be eligible to participate after a 1 month washout period.
* Use of PPI or H2R antagonist within 1 month of screening. The screened participant could be eligible to participate after a 1 month washout period.
* Daily use of non-steroidal anti-inflammatory drugs, cortisone, or other anti-inflammatory drugs 1 month prior to screening. The screened participant could be eligible to participate after a 1 month washout period.
* Current use, or use within the past 1 month, of narcotics or other medications for IBS symptom management (e.g. alosetron, tegaserod, lubiprostone, antispasmodics, antidiarrheals, laxatives, antipsychotics, tricyclic anti-depressants, selective serotonin reuptake inhibitors (SSRIs)). Subjects taking a stable dose of anti-depressants for at least 30 days with no plan to change dosage during the trial will be eligible for inclusion in the study.
* Regular use of anti-diarrhea medications and laxatives. Occasional use is permitted prior to screening (≤ than once a month); if current use is >once per month a one month wash out period is needed prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
IBS Symptom Severity Score | 8 Weeks
  Assessed using IBS Severity Scoring System Questionnaire, Part I.

SECONDARY OUTCOMES:
IBS Symptom Severity Score by IBS Subtype | 8 weeks
  Assessed using IBS Severity Scoring System Questionnaire, Part I.
Number of Responders | 8 weeks
  A responder is defined as a participant who has at least a 20% improvement in the IBS-SSS severity score after 8 weeks of supplementation
Anxiety and Depression | 8 weeks
  Assessed by administering the HADS questionnaire
Abdominal pain frequency | 8 weeks
  Assessed using IBS Severity Scoring System Questionnaire, Part I(c)
Abdominal distension/tightness | 8 weeks
  Assessed using the IBS-SSS Question 2(b)
Abdominal Pain Intensity | 8 weeks
  Mean weekly score. Assessed using IBS-SSS
Severity of straining | 8 weeks
  Assessed using IBS daily diary, 5 point ordinal scale
Health Status | 8 weeks
  Assessed by administration of the SF-36 questionnaire
Impact of IBS symptoms on Quality of Life | 8 weeks
  Assessed by administration of the IBS-QOL Questionnaire
Severity of IBS Symptoms | 4 weeks
  Assessed by administration of the IBS-SSS questionnaire, difference from baseline to week 4
Bowel Habit Satisfaction | 8 weeks
  Assessed by question 3 of the IBS-SSS
Stool Consistency | 8 weeks
  Assessed using the Bristol Stool Scale included in the IBS Daily Diary
Stool Frequency | 8 weeks
  Assessed using the IBS Daily Diary

OTHER OUTCOMES:
Compliance and Recovery of Probiotic strains | 8 weeks
  Monitored by qPCR of fecal samples
Microbiome Composition | 8 weeks
  Detected in fecal samples
Cysteine and serine-protease activity | 8 weeks
  Measured in stool samples
Amount of rescue medication used throughout the trial | 8 weeks
  Use of rescue medication (Bisacodyl 5mg tablet)
Safety Anthropometric Measurements | 8 weeks
  Blood pressure, Heart rate, Weight and BMI
Safety blood parameters | 8 weeks
  Complete blood count, electrolytes, markers of kidney and liver function
Number of Adverse Events occurring throughout the trial | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada